CLINICAL TRIAL: NCT02858739
Title: Polymer Free Biolimus Eluting Stent Implantation In All Comers Population: Analysis Of Dapt Cessation And Clinical Outcome After Biofreedom Stent Implantation
Brief Title: Biofreedom Stent in All Comer Population
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gennaro Sardella, Director of Cardiac Invasive Cardiology, University of Roma La Sapienza
Other Study IDs: SARDELLA RUDI FREE
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BIOFREEDOM STENT

SUMMARY:
AIM OF THE STUDY: The aim of the present registry is to investigate the procedural as well as the long-term clinical results in terms of safety and efficacy of the polymer-free DES technology in all comers patients with an indication to percutaneous coronary intervention.

PRIMARY SAFETY ENDPOINTS: the cumulative hierarchical incidence of major adverse cardiac events (MACCE) defined as: cardiac death, non-fatal myocardial infarction (MI), stroke and ARC-defined stent thrombosis (18) at any time point and bleeding defined according to BARC classification (19).

PRIMARY EFFICACY ENDPOINTS: clinically driven target lesion revascularization (TLR).

STUDY DESIGN: multicenter (presumably 10 centers across the Italian territory), prospective observational registry aiming to enroll a population of 1000 patients.

STUDY DURATION: We project 12 months for recruitment, 5 year follow-up duration after last patient in the registry.

CLINICAL FOLLOW-UP PLAN: 30 days, 3, 6, 9 months, 1 year, and then yearly up to 5 years after the index procedure.

PATIENTS SELECTION CRITERIA:

This is an "all comers" registry and patient who will be enrolled have to meet the sequent criteria:

* Patient must be at least 18 years of age at the time of signing the Informed Consent Form after Biofreedom placement.
* All "de novo" lesion subsets are included.
* Patient must agree to undergo all required follow-up visits and data collection.
* Patient must have indication to percutaneous coronary intervention following:

  * Stable angina or evidence of myocardial ischemia with stress echocardiography/ myocardial SPECT/exercise test, or
  * Unstable angina / non ST-elevation myocardial infarction
  * ST-elevation myocardial infarction with de novo culprit lesion.

EXCLUSION CRITERIA:

The exclusion criteria must follow the most recent IFU which may include but are not limited to the following:

* Known intolerance to any of the device components
* In-stent restenosis
* Woman with childbearing potential
* Age < 18y/o
* Inability to provide written informed consent

EFFICACY PARAMETERS: TLR and TVR up to 5-year follow-up.

SAFETY "PATIENT ORIENTED" PARAMETERS: all cause mortality, any myocardial infarction, Stent thrombosis based on the ARC classification, up to 5-year follow-up and bleeding occurrence according to BARC classification. Data on dual antiplatelet therapy use will also be collected and analyzed according to duration and cessation modalities.

Sample size justification: Being this an observational registry aiming at quantifying effect estimates without direct comparisons to other devices for coronary angioplasty, we relied on confidence interval profiling for sample size justification, without proceeding with formal power analysis. The main analysis will be an overall and comprehensive analysis and it will be planned the primary analytical approach of all-comers patients with coronary artery disease and indication to PCI. Accordingly, we computed that a target sample of 1000 patients will enable the computation of reasonably precise 95% confidence intervals. Specifically, assuming a 8% MACE rate at 1 year (in keeping with RUDY study and LEADERS FREE trial design), confidence intervals computed with the adjusted Wald method would be 7.1% to 9.6% for a 1000-patient sample (point estimate 80/1000 [8.0%]). Given that the registry aims to reflect real-world patients and practice, no prevision to limit or restrict patient enrollment is considered.

Analytical plan: Continuous endpoints will be summarized by presenting the total number of patients, mean, standard deviation, median, minimum, and maximum. Tabulation of categorical parameters will include counts and percentages. The outcomes will be summarized as both a discrete and a continuous variable using the method described above. Survival analysis will be performed with the Kaplan-Meier method. Statistical inference will be based on the computation of 95% confidence intervals using the adjusted Wald method. Additional analyses will involve key subgroups defined according to baseline, lesion, and procedural features, with statistical significance set at the 5% 2-tailed level. Specifically, Student t, Fisher exact, and log-rank tests will be used for such bivariate analyses, whereas multivariable linear regression, logistic regression, and Cox proportional hazard analyses will be used to adjust for confounders.

DETAILED DESCRIPTION:
1. INTRODUCTION

   The RUDI FREE REGISTRY on the polymer-free DES (BIOFREEDOM) for coronary artery disease is a investigator-initiated, prospective, multicenter registry of all-comers patients with an indication to percutaneous coronary intervention. This Registry will enroll 1000 patients in approximately 10 sites throughout the Italian territory where BIOFREEDOM has regulatory approval and is commercially available.
2. BACKGROUND INFORMATION

2.1 Coronary device evolution

In 1977 Andreas Grüntzig performed the first balloon coronary angioplasty, a revolutionary treatment that lead to the birth of a new specialty, "interventional cardiology". Since that pioneering procedure, extensive developments and advances culminated in percutaneous coronary intervention (PCI) being one of the most frequently performed invasive medical procedures in clinical practice today. Coronary stenting became widely implemented after the publication of the landmark BENESTENT trial and the STRESS both with evidence indicating that stenting is safe in the absence of anticoagulation therapy with the use of dual antiplatelet therapy (DAPT) and/or adequate stent deployment in order to avoid the stent thrombosis phenomenon. By 1999, coronary stenting was performed in 84.2% of PCI procedures ; however, despite their obvious advantages, there were associated problems and concerns. Most notably and in addition to the risk of thrombosis, an iatrogenic problem emerged in the form of in-stent neointimal hyperplasia . The dramatic reduction in restenosis rates, seen with the use of these DES compared with BMS , has been the major driving force behind the exponential growth of PCI as a treatment for patients with coronary artery disease (CAD). Even drug-eluting permanent metallic stents, however, have some short and long-term limitations: a still unclear duration of dual antiplatelet therapy which is strongly linked to the risk of stent thrombosis that, although infrequent, is a ominous event with poor prognosis. Durable polymers in first-generation of DES, triggering hypersensitivity reactions and chronic inflammation in the vessel layers, may indeed promote stent thrombosis. Therefore, in order to overcome these late undesirable effects by reducing arterial wall toxicity, new DES platforms with more biocompatible durable polymers, biodegradable polymers or polymer-free have been developed.

2.2 BIOFREEDOM technology

The Biolimus A9-coated BioFreedom is a drug-coated stent (DCS) that consists of a stainless steel stent platform with a textured abluminal surface onto which BA9 in solvent is applied . The drug-coated stent is crimped onto a delivery system which includes a high pressure, semi-compliant balloon incorporated onto the distal tip of a rapid exchange delivery catheter system. The delivery system has two radiopaque markers inside the balloon, which fluoroscopically mark the ends of the stent to facilitate proper stent placement. For this trial, the BioFreedom DCS will be available in 6 nominal stent diameters (2.25-4.0 mm), seven lengths (8-28 mm), and a dose of Biolimus A9 of 15.6 μg/mm of stent length. After implantation, the stent thus releases the anti-proliferative agent directly into the vessel wall, without the use of any polymer in the coating, thereby eliminating polymer associated tissue responses. BA9 is extremely lipophilic, and once it is taken up by the vessel wall, a process that is 98% complete at 4 weeks in an animal model, the stent becomes a BMS. In a pig model at 28 and 180 days, BioFreedom stents were associated with an inflammation score that was significantly lower than Cypher sirolimus eluting polymer-coated stents, and similar to that observed with BMS . It is therefore reasonable to hypothesize that this DCS may have a safety advantage, with a lesser dependence on prolonged DAPT than a polymer-associated DES. The anti-proliferative efficacy of the device was assessed in the BioFreedom first-in-man trial. Two different BA9 doses on the BioFreedom stent were compared to the Taxus Liberté stent in 182 low-risk patients, 92% of whom underwent control angiography at 4 or 12 months. DAPT was recommended for at least 6 months for all patients. The primary endpoint was a non-inferiority comparison between BioFreedom standard dose and Taxus of mean in-stent late lumen loss at 12 months (P = .001). In addition, median in-stent late loss was compared among the three groups in the study, resulting in values of 0.17 mm for the standard dose (15.6 μg/mm), 0.22 mm for the low dose (7.8 μg/mm), and 0.35 mm for the Taxus stent (standard dose vs Taxus: superiority P = .11). At 2 years clinically-driven target lesion revascularization (TLR) was 3.4% for the standard dose BioFreedom, 9.9% for the low dose and 5.0% for the Taxus (ns). There was no ST in any patient up to 2 years. Based on these results, the standard dose device was selected for further clinical evaluation. Recently has been published the rationale and design of the LEADERS FREE trial : A randomized double-blind comparison of the BioFreedom drug-coated stent vs the Gazelle bare metal stent in patients at high bleeding risk using a short (1 month) course of dual antiplatelet therapy. A total of 2456 patients considered at high risk of bleeding will be randomized in a double-blind fashion to the BioFreedom drug-coated stent or to a control arm (Gazelle bare metal stent). Both groups will be treated with DAPT during 1 month only, followed by long-term aspirin alone. At 1-year follow-up, the primary safety endpoint (a composite of cardiac death, myocardial infarction and stent thrombosis) will be assessed by a non-inferiority analysis, and the primary efficacy endpoint (clinically driven target lesion revascularization) by a superiority analysis. This trial should help better characterize a neglected subset of PCI patients and quantify both their thrombotic and bleeding risks.

2.2 STUDY DEVICE

The device to be used in this registry is the the Biolimus A9-coated BioFreedom stent (DCS) System manufactured by Biosensors. The Biofreedom stent refers to a system that consists of the drug-coated stent that is crimped onto a delivery system (see the IFU for details concerning indications for use, contraindications, system preparation, precautions, and warnings).

3 REGISTRY OBJECTIVE

The aim of the present registry is to investigate the procedural as well as the long-term clinical results in terms of safety and efficacy of the polymer-free DES technology in all comers patients with an indication to percutaneous coronary intervention.

4 REGISTRY FLOW AND CLINICAL FOLLOW-UP SCHEDULE

The RUDI FREE REGISTRY is a prospective multi-center national registry evaluating the safety and efficacy in terns of procedural and clinical outcomes of the BIOFREEDOM stent in daily use in all comers patients with indication to PCI. All lesion subsets are included. DAPT cessation will be left to operator's discretion according to the different clinical characteristics of the patients (high bleeding risk, stable and ACS population).

4.1 Number of Patients to be Registered and Patient Follow-up

The RUDI FREE REGISTRY will enroll approximately 1000 pts in about 10 sites throughout the Italian territory where Biofreedom stent has regulatory approval and is commercially available.

Patients will have clinical follow-up by telephone contact or office visits.

4.2 Measures Taken to Avoid and Minimize Bias

In order to minimize bias in assessing MACCE outcomes, these events will be adjudicated by an independent committee.

4.3 Clinical follow-up plan: 30 days, 3, 6 months, 1 year, and then yearly up to 5 years after the index procedure.

Angiographic follow-up will be performed ischemia driven 5. OUTCOMES/ENDPOINTS

Outcomes are as specified below:

5.1 Primary safety endpoints: the cumulative hierarchical incidence of major adverse cardiac events (MACCE) defined as: cardiac death, non-fatal myocardial infarction (MI), stroke and ARC-defined stent thrombosis at any time point and bleeding defined according to BARC classification.

5.2 Primary efficacy endpoints: clinically driven target lesion revascularization (TLR).

5.3 Efficacy parameters: TLR and TVR up to 5-year follow-up. 5.4 Safety "patient oriented" parameters: all cause mortality, any myocardial infarction, Stent thrombosis based on the ARC classification, up to 5-year follow-up. Data on dual antiplatelet therapy use will also be collected and analyzed according with the difference in terms of duration (according with operator's discretion) and cessation according with the new classification by PARIS study

6. PATIENTS

6.1 Patient Population

Patients enrolled into this registry will be male and female patients derived from the general interventional cardiology population who satisfy the inclusion and exclusion criteria. The RUDI FREE REGISTRY will enroll 1000 patients in approximately 10 sites throughout the national territory (see section 4.1).

6.2 Patient Screening and Informed Consent

6.2.1 Patient Screening All patients admitted for PCI with Biofreedom stent should be evaluated for participation in the registry.

6.2.2 Informed Consent

The Investigator or designee, who has been trained on the protocol, will explain the nature and scope of the registry and inform the patient of the potential risks and benefits of participation, and document consent to treatment with an Biofreedom stent according to standard hospital practice. For this registry the patient must consent to data collection and follow-up visits. All patients (or legally authorized patients' representatives if applicable) must sign, date and time Medical Ethics Committee (MEC) approved informed consent prior to data collection for this registry. Obtaining the consent, provision of a copy to the patient, along with the date and time must be documented in the patient's medical records. The informed consent form must be signed by the investigator. In addition, the signed informed consent must be kept in the patient's medical records.

6.3 Eligibility Criteria

6.3.1 General Eligibility Criteria

Patients enrolled into this registry will be male and female patients derived from the general interventional cardiology population who are scheduled for PCI and BIOFREEDOM implantation. All patients admitted for PCI should be evaluated for participation in the registry. The choice of this stent will be left to the operators' discretion considering the coronary anatomy, lesions characteristics, patients characteristics. Patients must meet the inclusion criteria to be considered for the registry. If any of the exclusion criteria is met, the patient will be excluded from the clinical evaluation and cannot be registered.

On the basis of patients characteristics the DAPT recommendation will be left to operator's discretion according with PCI guidelines and basal clinical patient's charachteristics in terms of high bleeding risk feature, stable and ACS patients Data on dual antiplatelet therapy use will also be collected and analyzed with a particular focus on different DAPT cessation (discontinuation, interruption and disruption) as defined in PARIS registry.

6.4 Patient Discontinuation

Once registered, each patient shall remain in the registry until completion of the required follow-up period; however, a patient's participation is voluntary and the patient has the right to withdraw at any time without penalty or loss of benefit. Conceivable reasons for discontinuation may include but not be limited to the following:

* Patient voluntary withdrawal
* Patient withdrawal by physician as clinically-indicated
* Patient lost-to-follow-up: If the patient misses two consecutive scheduled follow up time points, and attempts at contacting the patient are unsuccessful, then the patient is considered lost to follow-up.

No additional data is needed and will be recorded from patients once withdrawn from the registry. Patients will not be replaced.

6.5 Registry Completion

An eCRF registry completion form must be completed when:

* the patient is considered lost-to-follow-up per the above definition or
* the patient withdraws from the registry or
* the investigator withdraws the patient from the registry or
* the patient's follow-up is terminated upon registry follow-up completed (see Section 4.3 for details)

  7. TREATMENT AND SCHEDULE OF EVENTS

The treatment strategy will be determined by the investigator. It is required that each enrolling investigator review the most recent Biofreedom IFU and assess the contraindications, warnings and precaution sections with respect to the risks and benefits for treating potential patients.

7.1 Baseline

Patient preparation will be in accordance with standard hospital policy for the care of interventional cardiology patients.

Baseline data will be collected as per eCRF. The Syntax score will be calculated in all patients.

7.2 Procedure

During the procedure, patients will receive appropriate anticoagulation and other therapies according to standard hospital practice.

QCA analysis is recommended pre implantation of the BIOFREEDOM stent, for correct sizing. IVUS, VH-IVUS and OCT techniques are encouraged. These imaging tools will be subject of subgroup analysis.

7.3 Post-procedure (In-hospital)

Post procedure data will be collected as per eCRF

7.3.1 Follow-up Antiplatelet Medications

As informed previously minimum of 6 months duration of DAPT is recommended with variations left to operator's discretion according to the previous expressed clinica patient's charactreistics.. Specific type of DAPT will be recorded as per eCRF considering the new PARIS classification of DAPT cessation

7.4 Clinical Follow-up

• Clinical follow-up will be performed at 30 days, 3, 6 months, 1 year and then yearly up to 5 years after the index procedure: office visit is encouraged after the index procedure by telephone contact or office visits. Office visit will be encouraged. The angiographic follow up will be clinically driven.

7.5 Angiographic follow up

The angiographic follow up will be clinically driven. However, patients undergoing angio follow up and IVUS or OCT follow up will be included in subgroup analysis and judicated by internal observers.

8. ADJUDICATION OF EVENTS

In order to minimize bias in assessing MACCE outcomes, these events will be adjudicated by an independent Clinical Event Committee. A Data Safety and Monitoring Board will also be established.

9. STATISTICAL ANALYSIS

9.1 Statistical Overview

The data will be reviewed by a Data Safety and Monitoring Board.

The Data Safety and Monitoring Board will be also responsible for:

* Determining whether information collected are sufficient to address the objectives
* Recommending modifications to the statistical analysis plan to address additional research questions based on review of the data

9.2 Analysis Population

All patients who are successfully registered will be included in the analysis. 9.3 Sample Size Calculations and Assumptions

Being this an observational registry aiming at quantifying effect estimates without direct comparisons to other devices for coronary angioplasty, we relied on confidence interval profiling for sample size justification, without proceeding with formal power analysis. The main analysis will be an overall and comprehensive analysis and it will be planned the primary analytical approach of all-comers patients with coronary artery disease and indication to PCI. Accordingly, we computed that a target sample of 1000 patients will enable the computation of reasonably precise 95% confidence intervals. Specifically, assuming a 8.0% MACE rate at 1 year (in keeping with RUDI 2 study and LEADERS FREE , confidence intervals computed with the adjusted Wald method would be 7.1% to 9.6% for a 1000-patient sample (point estimate 80/1000 [8.0%]). Given that the registry aims to reflect real-world patients and practice, no prevision to limit or restrict patient enrollment is considered .

9.4 Statistical Analyses Continuous endpoints will be summarized by presenting the total number of patients, mean, standard deviation, median, minimum, and maximum. Tabulation of categorical parameters will include counts and percentages. The outcomes will be summarized as both a discrete and a continuous variable using the method described above. Survival analysis will be performed with the Kaplan-Meier method. Statistical inference will be based on the computation of 95% confidence intervals using the adjusted Wald method. Additional analyses will involve key subgroups defined according to baseline, lesion, and procedural features, with statistical significance set at the 5% 2-tailed level. Specifically, Student t, Fisher exact, and log-rank tests will be used for such bivariate analyses, whereas multivariable linear regression, logistic regression, and Cox proportional hazard analyses will be used to adjust for confounders.

10. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The investigator/institution will permit direct access to source data/documents in order for registry-related monitoring, audits, MEC review, and regulatory inspections to be performed.

As part of the informed consent, the investigator or designee will obtain permission for registry monitors or regulatory authorities to review, in confidence, any records identifying the patients in this registry.

11. QUALITY CONTROL AND QUALITY ASSURANCE

11.1 Protocol and Informed Consent Approval The Principal Investigator at each site must confirm and agree with the content of the protocol prior to participation in this registry. Also, the Principal Investigator will obtain written approval of the protocol, informed consent form, and other registry related documents from the MEC. In addition, the investigator will take actions necessary for ongoing registry approval at their site per established procedures of the MEC.

The investigator will advise the MEC of the progress of this registry on a regular basis until registry completion as required by the MEC.

The investigator will submit any amendments to the protocol as well as associated informed consent form changes and obtain written MEC approval prior to implementation as required by the MEC.

11.2 Monitoring

A monitoring plan will be established. Remote monitoring by the CRO and source documents analysis for events throughout the study period by an independent Event Committee, will be conducted to ensure compliance with the protocol and applicable regulatory requirements.

12. DATA HANDLING AND RECORD KEEPING

For the registry duration, the investigator will maintain complete and accurate documentation including but not limited to the following: medical records, registry progress records, laboratory reports, electronic case report forms, signed informed consent forms, device serial numbers for monitoring malfunctions, correspondence with the MEC and registry monitor/Sponsor, SAE reports, and information regarding patient discontinuation or registry completion.

12.1 Source Documentation

* Medical history/physical condition of the patient before involvement in the registry sufficient to verify protocol entry criteria
* Dated and signed notes on the day of entry into the registry referencing the sponsor, protocol number, patient ID number and a statement that informed consent was obtained
* Dated and signed notes from each patient visit
* Adverse events reported and their resolution including supporting documents such as discharge summaries, catheterization laboratory reports, ECGs, and lab results including documentation of site awareness of SAEs and of investigator device relationship assessment of AEs.
* Notes regarding Dual Anti Platelet Therapy medications taken during the registry
* (including start and stop dates)
* Patient's condition upon completion of or withdrawal from the registry
* Any other data required to substantiate data entered into the CRF

12.2 Electronic Case Report Form Completion

Primary data collection based on source-documented hospital and /or clinic chart reviews will be performed clearly and accurately by site personnel trained on the protocol and eCRF completion. eCRF data will be collected for all patients that are registered.

13. ETHICAL CONSIDERATION

13.1 Medical Ethics Committee Review Medical Ethics Committee (MEC) approval for the protocol and informed consent form /other written information provided to the patient will be obtained by the Principal Investigator at each investigational site prior to participation in this registry. No changes will be made to the protocol or informed consent form or other written information provided to the patient without appropriate approvals by the MEC.

Until the registry is completed, the Investigator will advise his/her MEC of the progress of this registry, per MEC requirements.

Further, any amendments to the protocol as well as associated informed consent form changes will be submitted to the MEC and written approval obtained prior to implementation, according to each institution's MEC requirements.

APPENDIX I: ABBREVIATIONS AND ACRONYMS

%DS: percent diameter stenosis AE: adverse event CABG: coronary artery bypass graft CE: Conformité Européene (EU) DAPT: Dual Anti Platelet Therapy DES: drug eluting stent eCRF: electronic Case Report Form GCP: Good Clinical Practice IFU: Instructions for Use MACCE: major adverse cardiac and cerebrovascular event MEC: medical ethics committee MI: myocardial infarction PCI: percutaneous coronary intervention SAE: serious adverse event TLR: target lesion revascularization TVR: target vessel revascularization

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age at the time of signing the Informed Consent after Biofreedom placement Form .
* All lesion subsets are included.
* Patient must agree to undergo all required follow-up visits and data collection.
* Patient must have indication to percutaneous coronary intervention following:

  * Stable angina or evidence of myocardial ischemia with stress echocardiography/ myocardial SPECT/exercise test, or
  * Unstable angina / non ST-elevation myocardial infarction
  * ST-elevation myocardial infarction with de novo culprit lesion.

Exclusion Criteria:

* Known intolerance to any of the device components
* In-stent restenosis
* Woman with childbearing potential
* Age < 18y/o
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pts with coronary disease all comers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
the cumulative hierarchical incidence of major adverse cardiac events (MACCE) ARC-defined stent thrombosis at any time point and bleeding defined according to BARC classification | 12 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No